CLINICAL TRIAL: NCT03065309
Title: Determination of Remifentanil's ED50 for Rapid Sequence Intubation Avoiding Bradycardia and Hypotension in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of Anesthesia department, Brasilia University Hospital
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: TCC-Lara-2017
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Bradycardia; Hypotension
MeSH Terms: conditions — Bradycardia; Hypotension | interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: Adaptative clinical trial, Dixon's Up-And-Down Method
Masking Description: Participant will receive propofol before induction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients will receive bolus dose of remifentanil before intubation
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — bolus dose

SUMMARY:
This study will find the median effective dose of remifentanil for rapid sequence intubation which avoids bradycardia and hypotension

DETAILED DESCRIPTION:
Remifentanil is becoming popular for rapid sequence intubation because it has a fast onset and ultra-short half-life.

Remifentanil a potent opioid associated to bradycardia and hypotension at high doses.

ELIGIBILITY:
Inclusion Criteria:

* Indication of anesthesia induction

Exclusion Criteria:

* Protocol violation
* Monitoring problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-25 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
hemodynamic stability during rapid sequence intubation | from anesthesia induction up to 5 minutes
  no bradycardia and no hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimarães, MSc, Study Director — Head of Anesthesiology
Locations (1):
- Hospital das Forças Armadas, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided